CLINICAL TRIAL: NCT06364293
Title: An Early Warning Model of Unfavorable Outcomes Following Endovascular Interventional Treatment of Intracranial Aneurysms Based on Medical Image Analysis and Deep Learning Algorithm
Brief Title: An Early Warning Model of Unfavorable Outcomes Following Endovascular Interventional Treatment of Intracranial Aneurysm
Status: Enrolling by invitation | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: KY2023-261-01
Record Dates: First submitted 2024-04-03; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Intracranial Aneurysm
Keywords: Unfavorable imaging outcome; artificial intelligent prediction model; Deep learning
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- the cohort with or without unfavorable imaging outcome: Cohorts will be divided into the favorable imaging outcome group and unfavorable imaging outcome group according to the interpretation of the imaging outcome of the postoperative follow-up of intravascular interventional therapy for intracranial aneurysms
  Interventions: Other: Observational design does not include interventional behavior.

INTERVENTIONS:
Other: Observational design does not include interventional behavior. — Observational design does not include interventional behavior.

SUMMARY:
Endovascular treatment has become one of the primary treatment methods for intracranial aneurysms. The unfavorable outcomes during follow-up included aneurysm recurrence and long-term incomplete-occlusion, which would bring a high risk of rebleeding and retreatment. Previous studies have tried to predict the outcomes of aneurysms following endovascular treatment based on aneurysm characteristics including morphology, embolization packing degree, etc, but the conclusion was inconsistent. Hemodynamics of aneurysms and parent artery played a greater role in predicting outcomes following endovascular treatments. Investigators also found that the outcomes were determined by many factors, in which the demography, clinical indicators, treatment methods, and material selection can not be ignored, and the mechanism of unfavorable imaging outcomes should be explored using large samples of clinical cases and numerous variable parameters. The pre-experiment of investigators confirmed that artificial intelligence technology can meet the calculation requirements for deep mining and analysis of large sample data. This study aims to use the deep learning model to identify relevant risk factors and weights, establish a stable and accurate prediction model, then incorporate the prospective study to verify the model. The results will be very helpful in accurately predicting the adverse outcomes such as recurrence and long-term non-occlusion after endovascular treatment and help to improve the therapeutic strategy and avoid risk factors. Besides, the occurrence of ischemic or hemorrhagic complications during follow-up may affect the final follow-up outcome, so the analysis was included as one of the outcome events to evaluate the prognosis after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of intracranial aneurysm；
* Endovascular intervention was performed；
* The age is more than 18 years and less than 80 years;
* At least one follow-up of imaging data must be digital subtraction angiography with a time interval of 12 months or more;
* The quality of image data can satisfy morphological measurement and hemodynamic calculation;
* The patient family members were informed and consented to participate in the study.

Exclusion Criteria:

* Dynamic aneurysms with cerebrovascular malformation;
* Dissecting, fusiform or thrombotic aneurysms;
* Follow-up images were not digital subtraction angiography or data quality can not meet the hydrodynamic analysis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included the patients undergoing intravascular interventional treatment of intracranial aneurysms.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Unfavorable imaging outcome | through study completion, an average of 1 year
  Unfavorable imaging outcome included the recurrence and long-term incomplete aneurysm occlusion. Any enlarged imaging of the residual portion of the aneurysm is considered a recurrence compared to immediate postoperative imaging. At the last DSA follow-up longer than 12 months, the aneurysm was not completely occluded, showing aneurysm residual portion and development (Raymond scale 3) and was judged to be long-term incomplete aneurysm occlusion.)

SECONDARY OUTCOMES:
Hemorrhagic or ischemic complication occurred during the follow-up | through study completion, an average of 1 year
  Ischemic or hemorrhagic complications occurred in patients with intracranial aneurysms during follow-up after endovascular therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided